CLINICAL TRIAL: NCT01759953
Title: Randomized Controlled Trial to Assess the Educational Efficacy of a Serious Game for Teaching Insulin Therapy to Primary Care Physicians
Brief Title: Educational Efficacy Assessment of a Serious Game to Teach Insulin Therapy to Primary Care Physicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Leandro Arthur Diehl, Assistant Professor, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: InsuOnline-01
Record Dates: First submitted 2012-12-21; First posted 2013-01-03 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Knowledge, Attitudes, Practice
Keywords: Diabetes Mellitus; Insulin; Video Games; Medical Education; Educational Technology; Continuing Medical Education
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Behavior; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- InsuOnline game (Active Comparator): Playing the InsuOnline game, on the web, in the player´s own time and rhythm, until its end, as already described previously.
  Interventions: Other: Game
- Traditional CME (Active Comparator): Traditional learning session as used for Continuing Medical Education, on insulin therapy, including a short lecture and a group discussion of the same clinical cases presented in the InsuOnline game
  Interventions: Other: Traditional CME

INTERVENTIONS:
Other: Game — InsuOnline game, on the web, in the player´s own time and rhythm
  Other Names: InsuOnline game; Serious game; Web-based game
  Arms: InsuOnline game
Other: Traditional CME — In-classroom traditional learning session about insulin therapy for diabetes, using a presential short lecture and a group discussion of the same clinical cases presented in the InsuOnline game
  Other Names: Classroom education; Onsite learning session; Lecture and clinical cases discussion
  Arms: Traditional CME

SUMMARY:
Background: Physicians´ lack of knowledge contributes to underuse of insulin and poor glycemic control in adults with diabetes mellitus (DM). Traditional continuing medical education have limited efficacy, so new approaches are required.

Objective: We report the design of a trial to assess the educational efficacy of InsuOnline©, a game for education of primary care physicians (PCPs) on initiation and adjustment of insulin for the treatment of DM, which was designed to be: a) educationally adequate; and b) self-motivating and attractive.

Methods: A multidisciplinary team, with endocrinologists, experts in medical education, and programmers, was assembled for design and development of InsuOnline©, a serious game which includes game elements and a well-defined, evidence-based curriculum of topics on insulin therapy. The first step of our study will be usability and playability tests, with PCPs and medical students, playing the game on a desktop. After that and further adjusts, we will perform an unblinded randomized controlled trial, with PCPs who work in the city of Londrina, to assess the educational validity of the game. A group of 64 PCPs will play InsuOnline© on the web, and the control group, of 64 PCPs, will underwent traditional teaching activities (lecture and group discussion). Knowledge on how to initiate and adjust insulin will be assessed by a web-based multiple-choice questionnaire, and attitudes regarding diabetes/insulin will be assessed by Diabetes Attitude Scale 3, at 3 time points: before, immediately after, and 6 months after the intervention. Subjects´ general impressions on the interventions will also be assessed by free-text questions. Software logs will be reviewed.

DETAILED DESCRIPTION:
Achieving and maintaining good glycemic control is the mainstay of treatment of diabetes mellitus (DM). Unfortunately, only 24% to 56% of patients with DM are within the goal of A1c <7%, in most countries.

Worldwide, according with public health trends, most diabetics are treated by primary care physicians (PCPs), but these professionals lack knowledge and confidence on several aspects of DM management, specially regarding insulin use. This contributes to the common problem known as clinical inertia ("the failure to advance therapy when indicated"), underuse of insulin, and poor glycemic control.

Continuing medical education (CME) on DM and insulin is often advocated as a solution to optimize the knowledge and the practice of PCPs; however, traditional CME activities (such as lectures and group discussions) have small and short-lasting efficacy. Thus, new educational methods are urgently required.

Objectives: To describe the design of a randomized controlled trial to assess if InsuOnline©, a PC serious game for teaching PCPs about initiation and adjustment of insulin in the treatment of DM, can be educationally effective.

Methods

Game Design A multidisciplinary team was assembled: clinical endocrinologists (LAD, RZE), experts in medical education (PAG, MLSGJ, ICMC) and software developers/game designers (JBA, RMS). The endocrinologists compiled a list of main topics (the "minimum curriculum" of the game) on insulin initiation and adjustment, for treatment of adults with DM, in the context of a primary health care setting.

Periodic team meetings were scheduled during the design and development phases, to review each step, correct problems, and make decisions for the following stages, in an iterative process. The group agreed that the game should be developed in a way to satisfy 2 basic conditions: a) to be educationally adequate; and b) to be self-motivating and attractive to the final users.

Level Design Sixteen diabetic patients were created, reflecting common clinical scenarios in actual primary health care clinical practice, each one corresponding to at least one of the topics of game´s minimum curriculum. Each patient is a game level. The patients/levels are disposed in an increasing complexity order. The player´s avatar must take decisions on which is the best therapeutic option to improve each patient´s glycemic control. Right decisions lead to progression to the next level.

Interaction Ways and Game Elements Players´ interaction with the game is made via mouse. Several ways of interaction and game elements were included along the game, to make it a pleasant experience and to maximize players´ intrinsic motivation. The player can read patients´s clinical charts, dialogue with them (choosing among a few options of "talks"), see their lab tests or fingertip glucose readings, review their physical exam, answer to "quiz challenges", solve puzzles, get "tips" from the mentor and from a nurse, and, finally, prescribe insulin. Sound track, score, visual and sound effects, patients' "mood" (the patient gets angry if the player makes too many errors), and between-levels animation scenes ("machinimas") were also included, to improve gaming experience and players´ motivation.

Pedagogical Elements Several pedagogical elements were included in the game, aiming for the best educational effects, based on principles of Adult Learning and Problem-Based Learning: motivation, goal-orientation, relevancy-orientation, self-pacing, timely and appropriate feedback, reinforcement of learning, informal environment, contextualisation, and practical ("hands-on") approach with active participation of the learner.

The game gives immediate feedback (given by the character of the "mentor"), comparing player's decisions with recommendations from clinical guidelines. Correct decisions lead to gaining points and progression in the game. At every step, the game offers additional learning resources: PDF-format help files (algorithms, summaries, clinical pearls), orientation from a "mentor" character, and links to bibliographic references. If the player fails to make the right choices, he can try the same level again.

Usability and Playability Evaluation The next step will be usability and playability assessment. For this, we will enroll 4 physicians who work in the city of Londrina (2 female and 2 male; 2 with gaming/computer previous experience and 2 without experience) and 4 undergraduate medical students from UEL (2 female and 2 male, with and without gaming experience), whom will play the game on a desktop, in a controlled environment (lab for usability tests), each participant alone in a single session. Usability data will be assessed using web-based System Usability Scale (SUS), as previously described by Brooke, and playability will be assessed by web-based Heuristic Evaluation for Playability (HEP), as described by Desurvire et al. The actions of the players will be recorded by the software for further analysis by the researchers (LAD, RMS). Further adjustments will be made in the game, according to responses obtained in this phase of the study.

Educational Efficacy Assessment After final adjustments in the game, guided by usability and playability assessments, the efficacy of InsuOnline© as an educational tool will be assessed in an unblinded randomized controlled trial. We will send a letter of invitation to all primary care physicians (PCPs) who work in the city of Londrina to participate in the study; if those PCPs do not fulfill our sample size, we will also invite PCPs from other cities of the state of Paraná (Brazil), such as Maringá, Curitiba, or São José dos Pinhais. The PCPs which are willing to participate in the study will be included and randomized at study entry, using a random number generator, to one of 2 groups. We will exclude clinical endocrinologists or diabetologists.

Physicians enrolled in the Group A will be exposed to InsuOnline©. They will be asked to play the game until its end, on the web (with an individual login), in their own time and rhythm. Physicians enrolled in the Group B will undertake a traditional (in-class) learning session, during one afternoon, composed by a short lecture and a group discussion of clinical cases which will be identical to the ones included in InsuOnline©. This traditional learning session will focus on the same teaching topics of the game, and it will be coordinated by a clinical endocrinologist not linked to the research team, in order to avoid potential biases. This endocrinologist will be previously trained by the researcher endocrinologists, and he will use didactic material prepared by our team.

We will evaluate subjects´ knowledge on insulin therapy using a web-based questionnaire, containing 10 to 20 multiple-choice questions. The questions will be clinical vignettes of diabetic patients who require initiation and/or adjustment of insulin; for each, the participant should choose the best option for achieving a better glycemic control, according to current guidelines. Questions regarding insulin therapy will be chosen from the American Diabetes Association Self-Assessment Program, Module 2 (Pharmacological Treatment of Hyperglycemia), translated to Portuguese, and adapted to be compatible with the game´s clinical scenarios and learning objectives. Participants´ attitudes regarding diabetes will also be assessed, by the application of web-based Diabetes Attitudes Scale, version 3 (DAS-3). The questionnaire and the DAS-3 will be answered by the participants in 3 time points: before the intervention (pre-test), immediately after the intervention (after-test), and 6 months after the intervention (late-test). The average of right answers will be presented and compared: a) in the different time points, within each group (intragroup), using analysis of variance (ANOVA); and b) between the two groups, at each time point (intergroup), using Student´s t test. A bicaudal significance level of 0.05 will be adopted. Data analysis will be done by intention-to-treat, with last observation carried forward, which means that all randomized participants´ data will be included in the final analysis.

A few Likert-scale and free-text questions will also be asked to the participants at the end of each intervention, in order to assess their general impressions about the intervention (mostly to assess if it was pleasant or enjoyable). Software-recorded data on player´s usage of the game will be analyzed to assess: number of logins, time spent on the game, etc. For the participants in Group A who does not finish the game, the reasons for early withdrawal will be collected by an online questionnaire. We will contact (by phone or e-mail) at least twice the participants who eventually do not fulfill the questionnaires.

In order to detect a minimum difference of 0.5 standard deviation on the average of right answers, with 80% of statistical power, at 5% of significance level, we will need to include 128 subjects in our study (64 in each group). We will enroll 160 subjects (80 in each group), in order to compensate for an expected 25% dropout rate.

Ethical Considerations Participation will be anonymous and voluntary, and all subjects will previously provide written informed consent, according to Brazilian Health Ministry´s regulations (see the informed consent form in the Appendix). The study protocol was approved by our local Research Ethics Committee (UEL, #051/2011 and #051/2012), and registered by UEL research board (Research Project #07471).

ELIGIBILITY:
Inclusion Criteria:

* Primary care physicians working in Londrina or other cities from the state of Paraná, Brazil

Exclusion Criteria:

* Clinical Endocrinologists
* Diabetologists
* Refuse to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Knowledge on insulin therapy for diabetes | In up to one year
  Average number of correct answers to a standardized web-based questionnaire on use of insulin for treatment of diabetes

SECONDARY OUTCOMES:
Attitudes regarding diabetes/insulin | In up to one year
  Average score on web-based Diabetes Attitude Score 3

OTHER OUTCOMES:
General impressions about the intervention | In up to one year
  Comments from the participants about how they enjoyed the educational experience, assessed by a few web-based Likert-scale and free-text questions
Usage data | In up to one year
  Review of game usage data, collected from software-generated logs for each player: time spent on the game, number of logins, etc.
Reasons for not finishing the game | In up to one year
  Main reasons for not finishing the game, for the participants who do not play the InsuOnline game until its end.

CONTACTS AND LOCATIONS:
Overall Officials: Leandro A Diehl, M.D., MsC, Principal Investigator — Universidade Estadual de Londrina; Pedro A Gordan, M.D., PhD, Study Director — Universidade Estadual de Londrina; Izabel CM Coelho, M.D., PhD, Study Chair — Faculdades Pequeno Príncipe
Locations (1):
- Hospital Universitário de Londrina, Londrina, Paraná, Brazil

REFERENCES:
- [Background] American Diabetes Association. Standards of medical care in diabetes--2012. Diabetes Care. 2012 Jan;35 Suppl 1(Suppl 1):S11-63. doi: 10.2337/dc12-s011. No abstract available. PMID 22187469
- [Background] Mendes AB, Fittipaldi JA, Neves RC, Chacra AR, Moreira ED Jr. Prevalence and correlates of inadequate glycaemic control: results from a nationwide survey in 6,671 adults with diabetes in Brazil. Acta Diabetol. 2010 Jun;47(2):137-45. doi: 10.1007/s00592-009-0138-z. Epub 2009 Aug 5. PMID 19655083
- [Background] Hayes RP, Fitzgerald JT, Jacober SJ. Primary care physician beliefs about insulin initiation in patients with type 2 diabetes. Int J Clin Pract. 2008 Jun;62(6):860-8. doi: 10.1111/j.1742-1241.2008.01742.x. Epub 2008 Apr 3. PMID 18393965
- [Background] Peyrot M, Rubin RR, Lauritzen T, Skovlund SE, Snoek FJ, Matthews DR, Landgraf R, Kleinebreil L; International DAWN Advisory Panel. Resistance to insulin therapy among patients and providers: results of the cross-national Diabetes Attitudes, Wishes, and Needs (DAWN) study. Diabetes Care. 2005 Nov;28(11):2673-9. doi: 10.2337/diacare.28.11.2673. PMID 16249538
- [Background] Lehmann ED. Interactive educational simulators in diabetes care. Med Inform (Lond). 1997 Jan-Mar;22(1):47-76. doi: 10.3109/14639239709089834. PMID 9183780
- [Background] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR; American Diabetes Association (ADA); European Association for the Study of Diabetes (EASD). Management of hyperglycemia in type 2 diabetes: a patient-centered approach: position statement of the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2012 Jun;35(6):1364-79. doi: 10.2337/dc12-0413. Epub 2012 Apr 19. No abstract available. PMID 22517736
- [Background] Lerario AC, Chacra AR, Pimazoni-Netto A, Malerbi D, Gross JL, Oliveira JE, Gomes MB, Santos RD, Fonseca RM, Betti R, Raduan R. Algorithm for the treatment of type 2 diabetes: a position statement of Brazilian Diabetes Society. Diabetol Metab Syndr. 2010 Jun 8;2(1):35. doi: 10.1186/1758-5996-2-35. PMID 20529311
- [Background] Akl EA, Sackett K, Pretorius R, Erdley S, Bhoopathi PS, Mustafa R, Schunemann HJ. Educational games for health professionals. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD006411. doi: 10.1002/14651858.CD006411.pub2. PMID 18254103
- [Derived] Diehl LA, Souza RM, Gordan PA, Esteves RZ, Coelho IC. InsuOnline, an Electronic Game for Medical Education on Insulin Therapy: A Randomized Controlled Trial With Primary Care Physicians. J Med Internet Res. 2017 Mar 9;19(3):e72. doi: 10.2196/jmir.6944. PMID 28279950
- [Derived] Diehl LA, Souza RM, Alves JB, Gordan PA, Esteves RZ, Jorge ML, Coelho IC. InsuOnline, a Serious Game to Teach Insulin Therapy to Primary Care Physicians: Design of the Game and a Randomized Controlled Trial for Educational Validation. JMIR Res Protoc. 2013 Jan 21;2(1):e5. doi: 10.2196/resprot.2431. PMID 23612462